CLINICAL TRIAL: NCT00368797
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Efficacy and Safety Study of NV1FGF in Patients With Severe Peripheral Artery Occlusive Disease.
Brief Title: Efficacy and Safety Study of NV1FGF in Patients With Severe Peripheral Artery Occlusive Disease
Acronym: TALISMAN 201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFI6143; NV1FGF-PM201
Record Dates: First submitted 2006-08-24; First posted 2006-08-25 (Estimated); Last update posted 2008-11-18 (Estimated); Status verified 2008-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Gene Therapy; PAOD; CLI
MeSH Terms: conditions — Peripheral Arterial Disease

INTERVENTIONS:
Drug: XRP0038 (NV1FGF)

SUMMARY:
This study is a double-blind study to evaluate the efficacy and safety of NV1FGF, a pCOR plasmid constructed by inserting the gene coding for the FGF compared to placebo in patients with severe Peripheral Arterial Occlusive Disease, Fontaine's stage IV. The efficacy was assessed by the complete healing of at least one ulcer in the treated limb, 25 week post-baseline and secondary by the rate of amputation and death.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with severe Peripheral Artery Occlusive Disease defined as Rutherford's Grade III, category 5 or 6, or Fontaine's stage IV.
* Trophic lesions with no signs of healing (no reduction in ulcer size or depth) for at least 2 weeks prior to first study treatment administration (Day 1).
* Patients with objective evidence of peripheral vascular disease (resting ankle pressure < 70 mmHg and/or toe pressure < 50 mmHg, and/or resting ankle-brachial index (ABI) < 0.4 and/or resting toe-brachial index (TBI) < 0.3 and/or metatarsal pulse volume recording (PVR) flat or barely pulsatile) in the diseased limb on two consecutive examinations performed at least 1 week apart.
* Demonstration or documentation (historical data not older than 6 months prior to first study treatment administration) of total occlusion of the affected limb of one or more of the iliac, superficial femoral, popliteal and/or one or more infrapopliteal arteries as assessed by angiography.
* Life expectancy > 6 months from the first study treatment administration.
* Poor/not candidates for revascularization (patients suitable for revascularization but with a high risk of failure/ amputation/ or patients not suitable for revascularization).

Exclusion Criteria:

* Previous or current history of malignant disease. Patients who had successful tumor resection or radio-chemotherapy more than 5 years prior to inclusion in the study and no recurrence will be allowed for inclusion.
* Suspicion of malignant disease (abnormal X ray,positive. stool hemoccult, positive Prostate Specific Antigen , abnormal mammography, papanicolaou smear of Class IV or Class V characterization.
* Lower extremity surgery : bypass/angioplasty of the leg to be treated within 2 months prior to the first administration of study treatment (Day 1).
* Active proliferative retinopathy.
* Buerger's disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2002-03; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Primary efficacy parameter: ulcer healing.
Ulcers will be evaluated at each visit primarily by collecting quantitative and qualitative information.

SECONDARY OUTCOMES:
Hemodynamic parameters:ABI, TcPO2
Pain
Amputation (Date of amputation, Indication for amputation, amputation level (minor and major)
Death

CONTACTS AND LOCATIONS:
Overall Officials: Sigrid NIKOL, Prof., Principal Investigator — Universitätsklinikum Münster
Locations (6):
- Ghent University Hospital, Ghent, Belgium
- Hôpital Européen Georges Pompidou, Paris, France
- Klinikum Karlsbad-Langensteinbach, Karlsbad, Germany
- Istituto Dermopatico dell'Immacolata, Roma, Italy
- Universitätsklinik, Bern, Switzerland
- St George's Hospital, London, United Kingdom

REFERENCES:
- [Result] Nikol S, Baumgartner I, Van Belle E, Diehm C, Visona A, Capogrossi MC, Ferreira-Maldent N, Gallino A, Wyatt MG, Wijesinghe LD, Fusari M, Stephan D, Emmerich J, Pompilio G, Vermassen F, Pham E, Grek V, Coleman M, Meyer F; TALISMAN 201 investigators. Therapeutic angiogenesis with intramuscular NV1FGF improves amputation-free survival in patients with critical limb ischemia. Mol Ther. 2008 May;16(5):972-8. doi: 10.1038/mt.2008.33. Epub 2008 Apr 1. PMID 18388929
- [Derived] Niebuhr A, Henry T, Goldman J, Baumgartner I, van Belle E, Gerss J, Hirsch AT, Nikol S. Long-term safety of intramuscular gene transfer of non-viral FGF1 for peripheral artery disease. Gene Ther. 2012 Mar;19(3):264-70. doi: 10.1038/gt.2011.85. Epub 2011 Jun 30. PMID 21716303
- See also: Related Info — http://www.sanofi-aventis.com